CLINICAL TRIAL: NCT00409591
Title: Maternal and Infant Peripartum Nevirapine, Versus Infant Only Peripartum Nevirapine, or Maternal Lopinavir/Ritonavir in Addition to Standard Zidovudine Prophylaxis for the Prevention of Perinatal HIV in Thailand.
Brief Title: Maternal/Infant Peripartum NVP, Versus Infant Only Peripartum NVP, or Maternal LPV/r in Addition to Standard ZDV Prophylaxis for the Prevention of Perinatal (PMTCT) HIV in Thailand
Acronym: PHPT-5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Change in National PMTCT guidelines in Thailand
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Harvard School of Public Health (HSPH) (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Marc Lallemant, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHPT-5 First Phase; R01HD052461 (NIH); R01HD056953 (NIH)
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections; Pregnancy
Keywords: Thailand; Developing Countries; Prophylaxis; Mother-to-child transmission; HIV-1; HIV-1 infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): NVP-NVP:
  * In women, one NVP 200 mg tablet at onset of labor;
  * In neonates, NVP oral suspension 6 mg in the delivery room immediately after birth plus a second dose between 48 and 72 hours
  Interventions: Drug: Maternal and infant nevirapine; Drug: zidovudine
- 2 (Experimental): PL-NVP:
  * In women, one placebo tablet at onset of labor;
  * In neonates, NVP oral suspension 6 mg in the delivery room immediately after birth plus a second dose between 48 and 72 hours
  Interventions: Drug: Maternal placebo and infant nevirapine; Drug: zidovudine
- 3 (Experimental): LPV/r:
  * In women, LPV/r 400/100 mg bid from 28 weeks' gestation until delivery
  Interventions: Drug: Maternal lopinavir+ritonavir; Drug: zidovudine

INTERVENTIONS:
Drug: Maternal and infant nevirapine — * In women, one NVP 200 mg tablet at onset of labor;
  * In neonates, NVP oral suspension 6 mg in the delivery room immediately
  Arms: 1
Drug: Maternal placebo and infant nevirapine — * In women, one placebo tablet at onset of labor;
  * In neonates, NVP oral suspension 6 mg in the delivery room immediately after birth plus a second dose between 48 and 72 hours
  Comparison between Arms 1 and 2 is double-blinded.
  Arms: 2
Drug: Maternal lopinavir+ritonavir — - In women, LPV/r 400/100 mg bid from 28 weeks' gestation until delivery
  Arms: 3
Drug: zidovudine — In addition, all women and infants in the 3 arms will receive standard ZDV prophylaxis, as per Thai and WHO guidelines.

SUMMARY:
The purpose of this study is to compare the efficacy of two doses of nevirapine (NVP) given only to the infants or lopinavir/ritonavir (LPV/r) from 28 weeks gestation with single dose (SD) NVP given to the mothers plus two doses to the infants, in addition to zidovudine (ZDV) prophylaxis (from 28 weeks' gestation and for one week of ZDV in neonates) for the prevention of mother-to-child transmission of HIV-1.

DETAILED DESCRIPTION:
Multicenter, placebo-controlled, double blind, clinical trial where non immunocompromised women receiving the ZDV prophylaxis regimen from 28 weeks gestation, as recommended in Thailand, will be randomized to one of two arms:

Arm 1: NVP-NVP:

* In women, one NVP 200 mg tablet at onset of labor+;
* In neonates, NVP oral suspension 6 mg in the delivery room immediately after birth plus a second dose between 48 and 72 hours+++

Arm 2: PL-NVP:

* In women, one placebo tablet at onset of labor++;
* In neonates, NVP oral suspension 6 mg in the delivery room immediately after birth plus a second dose between 48 and 72 hours+++

Arm 3: LPV/r:

* In women, LPV/r 400/100 mg bid from 28 weeks' gestation until delivery

  * women in Arm 1 will also receive 7-day ZDV 300mg bid plus 3TC 150mg bid from delivery. ++women in Arm 2 will also receive 7-day (ZDV+3TC) Placebo from delivery. +++If the new born weight less than 2500 g, nevirapine will be administered 2 mg./1 kg (As per Thai Guideline).

All infants will receive ZDV for at least one week. Follow-up of women and infants is carried out on an outpatient basis except for delivery and the first three days after delivery. Mothers and infants are followed-up for 24 months after delivery.

Note: The study was stopped and data unblinded upon DSMB recommendations in September 2010 because of changes in Thai PMTCT guidelines recommending use of HAART in all HIV infected pregnant women regardless of their CD4 count. At the time of unblinding 435 pregnant women had been enrolled and follow-up of these women and their children is continuing.

ELIGIBILITY:
Pre-Entry Criteria

* Evidence of HIV infection (documented by two HIV antibody tests on two different dates)
* Intend to be followed at a study site for the duration of the study
* At least 18 years old
* Written informed consent.

Inclusion Criteria:

Women are eligible for the study if they

* met all pre-entry criteria
* Evidence of HIV infection, as documented by two serology tests obtained at two different dates;
* between 28 and 36 weeks gestational age;
* antiretroviral naïve except for exposure to ZDV prophylaxis PMTCT;
* CD4 count above 250 cells/mm3 (within 4 months prior to randomization)
* agreement not to breastfeed;
* consent to participate and to be followed for the duration of the study;
* and the following laboratory values within 14 days prior to randomization:
* hemoglobin > 8.5 mg/dl;
* absolute neutrophil count > 750 cells/mm3;
* platelets > 50,000 cells/mm3;
* SGPT ≤ 5 times upper limit of normal;
* serum creatinine ≤ 1.5 times upper limit of normal (women with a serum creatinine > 1.5 times upper limit of normal must have a measured eight-hour urine creatinine clearance > 70 ml/min).

Exclusion criteria:

* Evidence of pre-existing fetal anomalies incompatible with life;
* patients who meet the criteria of Classes III/IV of the WHO classification of HIV-associated clinical disease;
* known hypersensitivity to any benzodiazepine;
* active tuberculosis;
* concurrent participation to any other clinical trial;
* receipt of benzodiazepines or antiretroviral agent other than ZDV;
* uncontrolled hypertension;
* anticoagulant therapy or magnesium sulfate within 2 weeks of enrollment or the need for them during labor or at delivery.

If any of these conditions occurs after randomization, the women will be excluded from study drug dosing. Women with CD4 count lower than 250 cells/mm3 will be excluded from the study and offered HAART in the context of the national program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Definitive HIV infection in infants as assessed by positive HIV DNA PCR on two peripheral blood samples | At birth, 7-10 days, 1, 2, 4 and 6 months of age

SECONDARY OUTCOMES:
Safety for mothers and children of two NVP doses in neonates with and without maternal single dose NVP at onset of labor or LPV/r from 28 weeks gestation. | From randomization during pregnancy until 24 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, MD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (43):
- Thailand (43):
  - Health Promotion Hospital Regional Center I, Bangkok, Bangkok
  - Nopparat Rajathanee Hospital, Kannayao, Bangkok
  - Bhumibol Adulyadej Hospital, Saimai, Bangkok
  - Chachoengsao Hospital, Muang, Changwat Chachoengsao
  - Prapokklao Hospital, Muang, Changwat Chanthaburi
  - Mae Chan Hospital, Mae Chan, Changwat Chiang Rai
  - Mae Sai Hospital, Mae Sai, Changwat Chiang Rai
  - Phan Hospital, Phan, Changwat Chiang Rai
  - Banglamung Hospital, Bang Lamung, Changwat Chon Buri
  - Somdej Pranangchao Sirikit Hospital, Chon Buri, Changwat Chon Buri
  - Chonburi Hospital, Muang, Changwat Chon Buri
  - Panasnikom Hospital, Panasnikom, Changwat Chon Buri
  - Ao Udom Hospital, Si Racha, Changwat Chon Buri
  - Kalasin Hospital, Muang, Changwat Kalasin
  - Regional Health Promotion Centre 6,, Khon Kaen, Changwat Khon Kaen
  - Khon Kaen Hospital, Muang, Changwat Khon Kaen
  - Lampang Hospital, Lampang, Changwat Lampang
  - Lamphun Hospital, Lamphun, Changwat Lamphun
  - Maharaj Nakhon Si Thammarat Hospital, Muang, Changwat Nakhon Si Thammarat
  - Nong Khai Hospital, Muang, Changwat Nong Khai
  - Pranangklao Hospital, Muang, Changwat Nonthaburi
  - Pathumthani Hospital, Muang, Changwat Pathum Thani
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Phayao Provincial Hospital, Phayao, Changwat Phayao
  - Buddhachinaraj Hospital, Muang, Changwat Phitsanulok
  - Rayong Hospital, Muang, Changwat Rayong
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Songkhla Hospital, Muangsongkhla, Changwat Songkhla
  - Trat Hospital, Muang, Changwat Trat
  - Health Promotion Center Region 10,, Chiang Mai, Chiang Mai
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - Sanpatong Hospital, Sanpatong, Chiang Mai
  - Chiang Saen Hospital, Chiang Saen, Chiangrai
  - Chiangrai Prachanukroh Hospital, Muang, Chiangrai
  - Wiangpapao Hospital, Wiangpapao, Chiangrai
  - Phaholpolphayuhasena Hospital, Munag, Kanchanaburi
  - Mahasarakam Hospital, Muang, Mahasarakam
  - Nakhonpathom Hospital, Muang, Nakhonpathom
  - Samutprakarn Hospital, Samutprakarn, Samutprakarn
  - Samutsakhon Hospital, Muang, Samutsakhon
  - Fang Hospital, Chiang Mai
  - Chomthong Hospital, Chiang Mai
  - Vachira Phuket Hospital, Phuket

REFERENCES:
- [Background] Lallemant M, Jourdain G, Le Coeur S, Mary JY, Ngo-Giang-Huong N, Koetsawang S, Kanshana S, McIntosh K, Thaineua V; Perinatal HIV Prevention Trial (Thailand) Investigators. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med. 2004 Jul 15;351(3):217-28. doi: 10.1056/NEJMoa033500. Epub 2004 Jul 9. PMID 15247338
- [Background] Jourdain G, Ngo-Giang-Huong N, Le Coeur S, Bowonwatanuwong C, Kantipong P, Leechanachai P, Ariyadej S, Leenasirimakul P, Hammer S, Lallemant M; Perinatal HIV Prevention Trial Group. Intrapartum exposure to nevirapine and subsequent maternal responses to nevirapine-based antiretroviral therapy. N Engl J Med. 2004 Jul 15;351(3):229-40. doi: 10.1056/NEJMoa041305. Epub 2004 Jul 9. PMID 15247339
- [Background] Shapiro RL, Thior I, Gilbert PB, Lockman S, Wester C, Smeaton LM, Stevens L, Heymann SJ, Ndung'u T, Gaseitsiwe S, Novitsky V, Makhema J, Lagakos S, Essex M. Maternal single-dose nevirapine versus placebo as part of an antiretroviral strategy to prevent mother-to-child HIV transmission in Botswana. AIDS. 2006 Jun 12;20(9):1281-8. doi: 10.1097/01.aids.0000232236.26630.35. PMID 16816557
- [Result] Cressey TR, Jourdain G, Rawangban B, Varadisai S, Kongpanichkul R, Sabsanong P, Yuthavisuthi P, Chirayus S, Ngo-Giang-Huong N, Voramongkol N, Pattarakulwanich S, Lallemant M; PHPT-5 Team. Pharmacokinetics and virologic response of zidovudine/lopinavir/ritonavir initiated during the third trimester of pregnancy. AIDS. 2010 Sep 10;24(14):2193-200. doi: 10.1097/QAD.0b013e32833ce57d. PMID 20625263
- [Result] Lallemant M, Le Coeur S, Sirirungsi W, Cressey TR, Ngo-Giang-Huong N, Traisathit P, Klinbuayaem V, Sabsanong P, Kanjanavikai P, Jourdain G, Mcintosh K, Koetsawang S; PHPT-5 study investigators. Randomized noninferiority trial of two maternal single-dose nevirapine-sparing regimens to prevent perinatal HIV in Thailand. AIDS. 2015 Nov 28;29(18):2497-507. doi: 10.1097/QAD.0000000000000865. PMID 26372485
- [Derived] Sripan P, Le Coeur S, Amzal B, Ingsrisawang L, Traisathit P, Ngo-Giang-Huong N, McIntosh K, Cressey TR, Sangsawang S, Rawangban B, Kanjanavikai P, Treluyer JM, Jourdain G, Lallemant M, Urien S. Modeling of In-Utero and Intra-Partum Transmissions to Evaluate the Efficacy of Interventions for the Prevention of Perinatal HIV. PLoS One. 2015 May 19;10(5):e0126647. doi: 10.1371/journal.pone.0126647. eCollection 2015. Erratum In: PLoS One. 2015 Jun 26;10(6):e0130917. doi: 10.1371/journal.pone.0130917. PLoS One. 2015 Aug 28;10(8):e0137368. doi: 10.1371/journal.pone.0137368. PMID 25992639
- See also: Program for HIV Prevention and Treatment (Thailand) — http://www.phpt.org